CLINICAL TRIAL: NCT06503081
Title: Investigating the Relationship Between Inflammation and Proteolytic Activity From Mucosa-associated Microbiota in Crohn's Disease Patients
Brief Title: Crohn's Disease - Inflammation and Microbial Proteolytic Activity
Acronym: CIMPA
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, David Armstrong, Professor of Medicine, McMaster University
Other Study IDs: HiREB-7789
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease of Both Small and Large Intestine
Keywords: Proteolytic activity; Serpin; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Crohn's disease: Patients previously diagnosed with Crohn's disease who have a clinical indication for undergoing a standard white light colonoscopy, as determined by their gastroenterologist, will be invited to participate. Patients undergoing colonoscopy for other indications (for example, for the investigation of possible malignancy, polyps, gastrointestinal bleeding or diarrhea, without colonic inflammation), will not be included in this study.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy with video recording and biopsy collection

SUMMARY:
This study postulates that altered microbiota associated with areas of mucosal inflammation in CD, can be characterized by an increased proteolytic profile. This is clinically important as it may be possible to modulate the proteolytic activity of the CD-associated bacteria by using other bacteria that produce protease inhibitors, such as serpins.

DETAILED DESCRIPTION:
Crohn's disease (CD), characterized by discontinuous intestinal injury and inflammation, has been associated with changes in the luminal microbiota and impaired barrier function. Previously, the investigators have shown that in patients with CD, the mucosa-associated microbiota is altered. Additionally, it has been shown that in patients with active CD, areas of intestinal injury are associated with impaired barrier function, but the mechanisms remain unclear. Increased host proteolytic activity has been reported in both CD and ulcerative colitis (UC). The microbiota is an important source of proteases with potential inflammatory and barrier disrupting capacity. Indeed, preliminary data indicate that in UC patients the gut microbiota contributes to proteolytic imbalance. It is unknown whether this is also the case in CD. Specifically, this study postulates that the altered microbiota associated with areas of mucosal inflammation in CD, is characterized by an increased proteolytic profile. This is clinically important as it may be possible to modulate the proteolytic activity of the CD-associated bacteria by using other bacteria that produce protease inhibitors such as serpins.

In this prospective observational study, patients booked for routine white light colonoscopy under the care of the Division of Gastroenterology, Hamilton Health Sciences at the McMaster University Medical Centre and Juravinski Hospital Endoscopy Units will be invited to participate. Patients previously diagnosed with Crohn's disease who have a clinical indication for undergoing a standard white light colonoscopy, as determined by the gastroenterologist, will be invited to participate; biopsy samples and mucosal brushings will be taken from inflamed and non-inflamed areas in the ileum or colon.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18 - 70 years old
* Have a confirmed diagnosis of Crohn's disease
* Have a clinical indication for standard, white light colonoscopy to assess disease activity and extent

Exclusion Criteria:

* Inability to provide written informed consent
* Presence of serious life-threatening co-morbidities
* Evidence of toxic megacolon, jaundice, cirrhosis, renal dysfunction, acute GI bleeding
* History of difficult colonoscopy, strictures or extensive diverticulosis
* Antibiotics in the last month
* Probiotics in the last week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be invited to participate in the outpatient clinic if the clinical need for standard, white light colonoscopy has already been confirmed as well as a previous diagnosis of Crohn's disease. All study subjects will be enrolled into the study after informed consent
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Altered microbiota associated with areas of mucosal inflammation in CD, is characterized by an increased proteolytic profile | December 2019 - January 2025
  Increase proteolytic activity profile influenced by microbiota composition in inflamed areas comprared with non-inflamed areas in a context of Crohn's disease

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Background] Bouma G, Strober W. The immunological and genetic basis of inflammatory bowel disease. Nat Rev Immunol. 2003 Jul;3(7):521-33. doi: 10.1038/nri1132. PMID 12876555
- [Background] Libertucci J, Dutta U, Kaur S, Jury J, Rossi L, Fontes ME, Shajib MS, Khan WI, Surette MG, Verdu EF, Armstrong D. Inflammation-related differences in mucosa-associated microbiota and intestinal barrier function in colonic Crohn's disease. Am J Physiol Gastrointest Liver Physiol. 2018 Sep 1;315(3):G420-G431. doi: 10.1152/ajpgi.00411.2017. Epub 2018 May 31. PMID 29848021
- [Background] Denadai-Souza A, Bonnart C, Tapias NS, Marcellin M, Gilmore B, Alric L, Bonnet D, Burlet-Schiltz O, Hollenberg MD, Vergnolle N, Deraison C. Functional Proteomic Profiling of Secreted Serine Proteases in Health and Inflammatory Bowel Disease. Sci Rep. 2018 May 18;8(1):7834. doi: 10.1038/s41598-018-26282-y. PMID 29777136
- [Background] Vergnolle N. Protease inhibition as new therapeutic strategy for GI diseases. Gut. 2016 Jul;65(7):1215-24. doi: 10.1136/gutjnl-2015-309147. Epub 2016 Apr 12. PMID 27196587
- [Background] Motta JP, Magne L, Descamps D, Rolland C, Squarzoni-Dale C, Rousset P, Martin L, Cenac N, Balloy V, Huerre M, Frohlich LF, Jenne D, Wartelle J, Belaaouaj A, Mas E, Vinel JP, Alric L, Chignard M, Vergnolle N, Sallenave JM. Modifying the protease, antiprotease pattern by elafin overexpression protects mice from colitis. Gastroenterology. 2011 Apr;140(4):1272-82. doi: 10.1053/j.gastro.2010.12.050. Epub 2011 Jan 1. PMID 21199654
- [Background] Caminero A, McCarville JL, Galipeau HJ, Deraison C, Bernier SP, Constante M, Rolland C, Meisel M, Murray JA, Yu XB, Alaedini A, Coombes BK, Bercik P, Southward CM, Ruf W, Jabri B, Chirdo FG, Casqueiro J, Surette MG, Vergnolle N, Verdu EF. Duodenal bacterial proteolytic activity determines sensitivity to dietary antigen through protease-activated receptor-2. Nat Commun. 2019 Mar 13;10(1):1198. doi: 10.1038/s41467-019-09037-9. PMID 30867416